CLINICAL TRIAL: NCT00978887
Title: Efficacy of Retorna Facial Cream Usage in the Treatment of Facial Wrinkles
Brief Title: Retorna Facial Cream in the Treatment of Facial Wrinkles
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Alfredo Abreu Daniel PhD, "Commander Manuel Fajardo Rivero" Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAT-0906-CU
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Facial Wrinkles
Keywords: Facial cream; natural product; facial wrinkles

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Retorna (facial cream)
  Interventions: Other: Retorna
- B (Placebo Comparator): Placebo (facial cream)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Retorna — Dosage commensurate with surface to be treated, Retorna facial cream (Topical use), twice a day, for 4 weeks.
  Arms: A
Other: Placebo — Dosage commensurate with surface to be treated, Placebo facial cream (Topical use), twice a day, for 4 weeks
  Arms: B

SUMMARY:
The purpose of the study is to assess the efficacy of Retorna facial cream usage in the reduction or total correction of facial wrinkles. The duration of this double-blind placebo controlled phase 3 clinical trial will be 4 weeks. The estimated number of women to be recruited and randomized for the study is 148. Occurrence of adverse effects will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Facial wrinkles
* Signed informed consent
* Given verbal agreement on solar exposure prevention within hours of intense solar radiation (10 am - 4 pm) by the usage of physical protection methods such as umbrellas, caps and hats.

Exclusion Criteria:

* Pregnancy
* Breast-feeding
* Use of steroids within 6 months.
* Patients under other experimental treatment
* Decompensated concomitant diseases
* Malignant neoplastic conditions.
* Alcoholism
* Handicap and/or psychiatric condition preventing treatment accomplishment.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 148 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Total correction or improvement of facial wrinkles at the end of treatment (4 weeks) | 4 weeks

SECONDARY OUTCOMES:
Presence of adverse effects within the 4 week treatment period | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose Dominguez Gómez, MD, Principal Investigator — "Commander Manuel Fajardo Rivero" Hospital
Locations (1):
- "Commander Manuel Fajardo Rivero" Hospital, Havana, La Habana, Cuba